CLINICAL TRIAL: NCT03335163
Title: The Effect of Topiramate on Etonogestrel Concentrations in Contraceptive Implant Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-1047
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Results first posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Migraine; Migraine;Menstrual; Contraception
MeSH Terms: conditions — Migraine Disorders | interventions — Topiramate

STUDY DESIGN:
Intervention Model Description: Prospective, non-inferiority study to evaluate the pharmacokinetic effect of topiramate on serum ENG levels in contraceptive implant users
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ENG Implant Users (Experimental): Healthy women using an ENG implant for at least 12 months and no greater than 36 months will be administered a 6 week titration schedule of topiramate to a max dose of 200mg bid by the final week.
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — Topiramate - Participants will undergo a 6 week titrated regimen of oral topiramate to reach a maximum dose of 400mg per day:
  Week 1 - topiramate PO 25mg daily Week 2 - topiramate PO 25mg twice daily Week 3 - topiramate PO 50mg twice daily Week 4 - topiramate PO 100mg twice daily Week 5 - topiramate PO 150mg twice daily Week 6 - topiramate PO 200mg twice daily

SUMMARY:
A prospective, non-inferiority study to evaluate the pharmacokinetic effect of topiramate on serum Etonogestrel (ENG) levels in contraceptive implant users.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, who have had an ENG implant for 12-36 months at the time of enrollment;
* Will maintain their implant during the study without modifications.

Exclusion Criteria:

* Women who are taking any medications or supplements known to be

  1. Cytochrome P-450 enzyme inducers, inhibitors, or substrates, and
  2. are not willing to abstain from any of these medications or supplements during the entire course of the study.
* Women with liver disease (i.e. hepatitis, fatty liver disease), and
* Women with abnormal liver or renal function, or
* Women with abnormal electrolytes on their screening blood work.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must have an ENG implant contraception method in place prior to entry into the study.
Enrollment: 48 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Teal, MD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lazorwitz A, Pena M, Sheeder J, Teal S. Effect of Topiramate on Serum Etonogestrel Concentrations Among Contraceptive Implant Users. Obstet Gynecol. 2022 Apr 1;139(4):579-587. doi: 10.1097/AOG.0000000000004697. Epub 2022 Mar 10. PMID 35594123

RESULTS

PARTICIPANT FLOW:
Groups:
- ENG Implant Users: Healthy women using an ENG implant for at least 12 months and no greater than 36 months will be administered a 6 week titration schedule of topiramate to a max dose of 200mg bid by the final week.
  Topiramate: Topiramate - Participants will undergo a 6 week titrated regimen of oral topiramate to reach a maximum dose of 400mg per day:
  Week 1 - topiramate PO 25mg daily Week 2 - topiramate PO 25mg twice daily Week 3 - topiramate PO 50mg twice daily Week 4 - topiramate PO 100mg twice daily Week 5 - topiramate PO 150mg twice daily Week 6 - topiramate PO 200mg twice daily
Period: Overall Study
Arm/Group | ENG Implant Users
Started | 48
Completed Visit 2 | 32
Completed Visit 3 | 31
Completed (Visit 4 completed) | 27
Not Completed | 21
Not completed — Not eligible due to laboratory criteria | 3
Not completed — Withdrawal by Subject | 18

BASELINE CHARACTERISTICS:
Population: Participants who completed at least one follow up visit
Arm/Group | ENG Implant Users
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 25.3 [18.3 to 37.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 23
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 32
Body-mass index [Median (Full Range); unit: kg/m^2] | 25.5 [18.7 to 42.2]
Duration of implant use [Median (Full Range); unit: months] | 24 [12 to 36]

OUTCOME MEASURES:

1. Primary Outcome: Serum Etonogestrel Concentrations
Description: The investigators will collect serum from participants at enrollment and at each of the three study follow-up visits. All samples will be batched for analysis. Analysis will be performed using a liquid-chromatography mass-spectrometry validated assay for measurement of serum etonogestrel concentration.
Time Frame: Enrollment (Baseline), 4 weeks (Visit 2), 5 weeks (Visit 3), 6 weeks (Visit 4)
Population: Due to early discontinuation from the study, data are available for only 31 participants for Visit 3 and 27 participants for Visit 4.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | ENG Implant Users
Number analyzed (Participants) | 32
pg/mL
  Baseline | 142.0 [76.2 to 771.0]
  Visit 2 | 126.0 [72.4 to 585.0]
  Visit 3: number analyzed (Participants) | 31
  Visit 3 | 119.0 [65.6 to 542.0]
  Visit 4: number analyzed (Participants) | 27
  Visit 4 | 105.0 [46.2 to 859.0]

ADVERSE EVENTS:
Time Frame: 11 weeks
Arm/Group | ENG Implant Users
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT03335163/Prot_SAP_000.pdf